CLINICAL TRIAL: NCT00368511
Title: The Nolwenn Effect in Geriatric Nursing Homes in the Netherlands
Brief Title: Fall Prevention Strategies Including Music and Posturography
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Carrick Institute for Graduate Studies (Other)
Responsible Party: Dr Roland Blaauw, Carrick Institute for Graduate Studies
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: CI-09-06-01
Record Dates: First submitted 2006-08-23; First posted 2006-08-24 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2008-05

CONDITIONS: Fall Prevention
Keywords: Fall Prevention; Dynamic Posturography; Nolwenn Effect; Music Listening

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (No Intervention): Listening to music and posture changes
  Interventions: Procedure: Music Listening

INTERVENTIONS:
Procedure: Music Listening — Listen to music and posture measurements

SUMMARY:
We propose to obtain computerized dynamic posturography scores on patients in a (psycho)geriatric nursing home utilizing the CAPS system from Vestibular Technology. This instrument has been validated to measure human stability and is associated with a Fall Probability percentage. Subjects will be asked to stand on a platform with eyes open and closed for approximately 30 seconds. The data obtained will be utilized as a base for change which can be compared to an outcome of music listening and fall prevention. Previous investigations have demonstrated a decrease in fall rates associated with music listening. We would like to measure the changes in human stability associated with a potential decrease in fall rates. We would also like to use the history of falls of the tested individuals if available. In case fall statistics are available we respectfully request access to all falls data available from the involved geriatric nursing home . The falls data will be kept confidential and only used as a control statistic in our evaluation of fall rates after implementation of our applications. The music used will include Nolwenn Leroy, Mozart and other Dutch and French Singers.

DETAILED DESCRIPTION:
The outcome measurement will be obtained using computerized dynamic posturography, a standard diagnostic test of balance function. The subject's balance will be tested using a three-component force platform (BalanceTRAK® CAPST - Vestibular Technologies, Cheyenne WY, USA) under one sensory condition of the modified Clinical Test of Sensory Interaction on Balance (mCTSIB), the eyes closed on perturbing surface condition. This condition was chosen as studies have shown it to be the single test that best correlates with balance impairment and falls. The stability score, already used in several studies by other authors will be used as the primary outcome measure in this research. It is defined as 1 minus the ratio between the measured sway during the test (computed as the major axis of a standard 95% confidence ellipse) and the amount of sway a normal subject of the same height as the one being tested should be able to sway before falling (also known as the theoretical maximum sway or the theoretical limit of stability, calculated using a regression formula based on the subject's height developed by NASA in 1962 and commonly used in all posturographic tests). For convenience, the stability score is expressed as a percentage. Its definition makes it a convenient and easy to understand measure to use as a subject able to stand perfectly still with no sway will have a score of 100%, whereas one that sways as much as the limit of stability will have a score of 0%. During each test, the subject's sway will be determined by the force platform and its related software. The CAPST three-component force platform uses 3 load cells arranged in a triangle to measure the distribution of the vertical ground reaction force on the platform. The analog load cell signals are amplified and simultaneously sampled by the platform electronics using three synchronized individual 24bit delta-sigma analog to digital converters sampling at 312kHz and decimating the samples to a data rate of 64Hz. The use of three A/D converters insures that the signals from the 3 load cells are acquired simultaneously with no timing error. The high sampling rate with the high decimation and low data rate of the sigma-delta converters eliminates aliasing and provides a resolution of about 4 parts per million. The digital load cell data will be sent via a USB connection to the PC where software uses a calibration matrix determined by the manufacturer to compute the total vertical force and the two horizontal moments acting on the platform. From these data, the software will compute the point of application of the vertical force acting on the platform, commonly referred to as the Center of Pressure (CoP). The location of the CoP coincides in static conditions with the projection of the subject's Center of Mass (CoM) onto the platform, and its movement relates to the movements of the subject's CoM (sway). The determination of the actual sway required the determination of the instantaneous location of the CoM will require the determination of the location and inertial properties of each body segment of the specific subject being tested. The CAPST, like every other posturographic equipment, uses the movement of the CoP as an approximation of the sway. Because it is an approximation, and because for kinetic reasons the CoP moves more than the CoM, the 95% confidence interval of the CoP motion will be considered. This will allow the CAPST software to compute the ellipse that represents the location of all of the sway samples collected during the test with 95% confidence. The major axis of this ellipse represents the maximum sway of the subject in any direction during the test and it is used to compute the stability score. To assess the accuracy and resolution of the measurement chain, calibrated weights of 75kg and 100kg will be positioned in the center of the force platform (as if it were a subject) and 20s acquisitions will be performed: the accuracy of the weight will be calibrated to fall within the instrument's factory specifications (+-2N). Therefore the accuracy for the position claimed by the manufacturer of +-1mm for a weight of 75kg will be accepted as correct as determination would require specialized equipment and software available only to the manufacturer. It should be noted that the overall accuracy of the position of the CoP given by the instrument will not be relevant in this study as the sway is determined by the motion of the CoP. The sway measurement error will be estimated considering the fact that during the test at both weights the dead weight will not move, but the measurement chain will indicate a "sway" of less then 0.05mm (measurement noise), therefore the resolution of the measurement chain and the sway measurement error will be considered to be 0.05mm. To verify the repeatability of the measurement chain, the same type of tests will be repeated two times, obtaining similar results (within the specified accuracy and resolution). Given the sway measurement error, the measurement error in the stability score will be determined. From the definition of the stability score it is clear that the least the theoretical limit of stability, the more pronounced the effect of the sway measurement error is. As the theoretical limit of stability is computed by using the formula 0.55*height*2*sin(6.25°), the shorter the subject, the more the stability score is sensitive to the measurement errors. To estimate the stability score measurement error a subject's height of 1.6m will be considered. Such a subject would have a theoretical limit of stability of 191.6mm. For such a subject, a sway measurement error of 0.05mm means a stability score measurement error of 0.05/191.6 or, if the score is expressed in percentage, of 0.026%. Thus, any changes in the stability score greater than that will be as a consequence of the subject's sway and not of measurement errors. Inpatients in Dutch Geriatric Hospitals will be randomized into several groups and all will have CAPS tests obtained. The groups will be asked to listen to a music specific song each morning and CAPS tests will be obtained after the listening experiences and at one month intervals throughout the study. Fall data will be collected as well and compared to previous falls data. The changes in CAPS outcomes as a measure of brain based postural change will be compared to normative data and the types of music listened to.

ELIGIBILITY:
Inclusion Criteria:

* Must be a full time in patient in a geriatric hospital in Holland

Exclusion Criteria:

* All others

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-08; Primary Completion 2007-03 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Historical Falls Data | Historical

CONTACTS AND LOCATIONS:
Overall Officials: Roland Blaauw, DC, DABCN, Study Director — Carrick Institute for Graduate Studies; Arjan Kuipers, DC, DABCN, Principal Investigator — Carrick Institute for Graduate Studies; Marko Blanker, MD, PhD, Principal Investigator — Carrick Institute for Graduate Studies; Frederick Carrick, PhD, FACCN, FICC, Study Chair — Carrick Institute for Graduate Studies
Locations (1):
- Carrick Institute for Graduate Studies-Gouda Netherlands, Gouda, Netherlands